CLINICAL TRIAL: NCT02447133
Title: TopQ Cut-off Score Validation Study for 3D OCT-1 Maestro
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Topcon 001-2015
Record Dates: First submitted 2015-05-11; First posted 2015-05-18 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Subjects Presenting With Normal Eyes
Keywords: no known ocular pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects Presenting With Normal Eyes: Subjects with no known ocular diseases will be scanned on the Maestro device
  Interventions: Device: 3D OCT-1 Maestro

INTERVENTIONS:
Device: 3D OCT-1 Maestro — OCT Machine used for diagnostic purposes

SUMMARY:
The objective of this study is to validate the TopQ cutoff scores, which have been previously determined.

DETAILED DESCRIPTION:
Scans with a TopQ score below the optimum cut-off should be considered to be poor or unacceptable quality, and scans with a TopQ score above the cut-off should be considered good or acceptable quality. The study will evaluate the predetermined cut-off values by investigating measurement variability of scans.

ELIGIBILITY:
Inclusion Criteria

1. Participants must be at least 18 years of age
2. They must be able to complete all testing (all OCT scans)
3. They must volunteer to be in the study and sign the consent form

Exclusion Criteria

1. Subject with history of ocular disease or ocular pathology
2. TopQ score from baseline OCT scan (i.e., without any ND filters) is below the cut-off value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with no known eye disease
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Sun, MD, Principal Investigator — Topcon Corporation
Locations (1):
- Topcon Medical Systems, Inc., Oakland, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Presenting With Normal Eyes
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Normal healthy eyes without any known eye conditions
Arm/Group | Subjects Presenting With Normal Eyes
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.17 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: TopQ Cut Off
Description: To validate the values of the predetermined TopQ score by showing the variability above and below the TopQ score of 25 for 12x9 Wide, 28 for 6x6 Macula, and 30 for 6x6 Disc scans.
Time Frame: 1 hour
Population: use of 12 subjects for 3 different scan patterns
Measure: Number; unit: microns
Groups:
- 12x9 Wide Scan: TopQ of 12x9 Wide Scan
- 6x6 Macula Scan: TopQ of 6x6 Macular Scan
- 6x6 Disc Scan: TopQ of 6x6 Disc Scan
Arm/Group | 12x9 Wide Scan | 6x6 Macula Scan | 6x6 Disc Scan
Number analyzed (Participants) | 12 | 12 | 12
microns
  Standard Deviation Above Threshold | 2.94 | 1.5 | 2.14
  Standard Deviation Below Threshold | 17.54 | 13.67 | 13.67

ADVERSE EVENTS:
Arm/Group | Subjects Presenting With Normal Eyes
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes